CLINICAL TRIAL: NCT03172689
Title: Validation of an Ultrasound Oesophageal Doppler Cardiac Output Monitor (ODM+, CardioQ) Versus a Transpulmonary Thermodilution Cardiac Output Monitor (TPTD, PiCCO)
Brief Title: Validation of CardioQ Versus PiCCO in Children
Acronym: CQPiCCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL57824.091.16
Record Dates: First submitted 2017-01-27; First posted 2017-06-01 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-11

CONDITIONS: Cardiac Output

STUDY DESIGN:
Intervention Model Description: children with an clinical indication for cardiac output monitoring in ICU or OR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CardioQ (Other): CardioQ will be used as CO monitor simultaneously with the standard of care PiCCO CO monitor
  Interventions: Device: CardioQ

INTERVENTIONS:
Device: CardioQ — comparison of cardiac output measurements between gold standard transpulmonary thermodilution (by PiCCO) versus an oesophageal doppler monitor (CardioQ) They will be used simultaneously
  Other Names: PiCCO

SUMMARY:
To compare the less invasive Oesophageal Doppler cardiac output Monitor (ODM) to the invasive (standard of care) Transpulmonary Thermodilution cardiac output monitor (TPTD) in children.

DETAILED DESCRIPTION:
This is a validation study. The study period starts as soon as CMO approval is acquired and will end after inclusion of 17 patients. This study is designed to test the effectiveness of a non invasive ODM catheter compared to the invasive, gold standard, TPTD technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0 to 16 years with an indication for invasive CO monitoring (TPTD). Indication for invasive CO monitoring always implies intubation and sedation.
* Signed informed consent

Exclusion Criteria:

* Congenital or acquired cardiovascular diseases (intracardiac/extracardiac intrathoracic shunt
* Cardiac valve diseases
* Aortic arch anomalies
* Tissue necrosis of oesophagus
* Carcinoma of pharynx, larynx of oesophagus
* Severe bleeding diatheses
* Age > 16 years
* Weight < 3.5 kg or > 50 kg.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Estimated)
Dates: Start 2017-08-29 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
cardiac output | 24 hours
  liter/m2/minute
stroke volume | 24 hours
  milliliters

SECONDARY OUTCOMES:
flow time corrected | 24 hours
  seconds
stroke distance | 24 hours
  centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Gert Jan Scheffer, prof. dr, Study Chair — Radboud University Medical Center
Locations (1):
- Radboud Univeristy Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No